CLINICAL TRIAL: NCT04096573
Title: A Phase 2, Multi Center, Randomized, Placebo Controlled Parallel Group Study to Evaluate the Clinical Efficacy and Safety of LC51 0255 in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: Efficacy and Safety of LC51-0255 in Subjects With Ulcerative Colitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: company decision
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-SGCL002
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LC51-0255 low dose (Experimental): Oral, daily, low dose for induction period, high dose for OLE period
  Interventions: Drug: LC51-0255
- LC51-0255 middle dose (Experimental): Oral, daily, middle dose for induction period, high dose for OLE period
  Interventions: Drug: LC51-0255
- LC51-0255 high dose (Experimental): Oral, daily, high dose for induction period, high dose for OLE period
  Interventions: Drug: LC51-0255
- placebo (Placebo Comparator): Oral, daily, placebo for induction period, high dose for OLE period
  Interventions: Drug: LC51-0255; Drug: Placebo

INTERVENTIONS:
Drug: LC51-0255 — LC51-0255
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
This is a Phase 2, multi center, randomized, placebo controlled parallel group study to evaluate the clinical efficacy and safety of LC51 0255 in subjects with moderately to severely active ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years
* Active UC confirmed by endoscopy
* Moderately to severely active UC defined as a 3-component Mayo Clinic score

Exclusion Criteria:

* Severe extensive colitis
* Diagnosis of microscopic colitis, ischemic colitis, or infectious colitis
* Treatment with cyclosporine, tacrolimus, sirolimus, methotrexate, or mycophenolate mofetil within 16 weeks of screening
* Treatment with a biologic agent (ie, anti TNFs, anti integrins, and anti interleukin 23) within 8 weeks prior to screening endoscopy
* Any prior exposure to S1P receptor modulators, natalizumab, lymphocyte-depleting therapies (ie, alemtuzumab, anti CD4, cladribine, rituximab, ocrelizumab, cyclophosphamide, mitoxantrone, total body irradiation, bone marrow transplantation, alemtuzumab, daclizumab)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | Week 12
  The proportion of subjects in clinical remission assessed by Mayo component sub-scores

SECONDARY OUTCOMES:
Clinical response | Week 12
  The proportion of subjects in clinical response assessed by Mayo component sub-scores
Endoscopic improvement and remission | Week 12
  The proportion of subjects in endoscopic improvement and remission assessed by Mayo endoscopic sub-score

OTHER OUTCOMES:
Clinical response and remission | Week 52
  The proportion of subjects in clinical response and remission assessed by Mayo component sub-scores
Endoscopic improvement and remission | Week 52
  The proportion of subjects in endoscopic improvement and remission assessed by Mayo endoscopic sub-score

IPD SHARING:
Plan to Share IPD: Undecided